CLINICAL TRIAL: NCT05301387
Title: The Effect of Ganglion Sphenopalatine Block (GSP-block) Versus Placebo on Postdural Puncture Headache: Follow Up
Brief Title: The Effect of Ganglion Sphenopalatine Block (GSP-block) Follow-Up
Acronym: GSP-FOLLOW
Status: Completed | Type: Observational
Sponsor: University Hospital Bispebjerg and Frederiksberg (Other)
Responsible Party: Principal Investigator, Mads Seit Jespersen, Principal Investigator, University Hospital Bispebjerg and Frederiksberg
Other Study IDs: GSPB-2018-FOLLOW
Record Dates: First submitted 2021-11-25; First posted 2022-03-29 (Actual); Last update posted 2022-04-29 (Actual); Status verified 2022-04

CONDITIONS: Post-Dural Puncture Headache; Ganglion Sphenopalatine Block
MeSH Terms: conditions — Post-Dural Puncture Headache | interventions — Sphenopalatine Ganglion Block

STUDY DESIGN:
Observational Model: Other | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Procedure: Ganglion Sphenopalatine Block — Block performed with bilaterally inserted q-tips with 1:1 mixture of lidocaine 40mg/ml and ropivacaine 5mg/mL or Block performed with bilaterally inserted q-tips with isotone NaCl

SUMMARY:
The purpose of this study is to evaluate the long term effects of the ganglion sphenopalatine block (GSP block) on postdural puncture headache.

DETAILED DESCRIPTION:
Adult patients with postdural puncture headache was enrolled in main study (NCT03652714). In the main study the patients was randomised to receive a ganglion sphenopalatine block (GSP-block) with either local anesthetic (lidocaine + ropivacaine) or placebo (isotone NaCl).

Following inclusion in the main study all participants are sent a follow-up questionnaire.

Primary outcome is disability due to headache defined as moderate to severe disability measured with Migraine Disability Assessment Test (MIDAS) in the 3 months following initial block and average pain score in the 3 months following the initial block on a 0-10 pain intensity scale.

Secondary outcome is disability due to headache defined as moderate to severe disability measured with Migraine Disability Assessment Test (MIDAS) in the 3 previous months as well as average pain scores in the previous 3 months, days with headache and long and short term side effects of the block.

ELIGIBILITY:
Patients who where included in main study and had the following eligibility criteria:

Inclusion Criteria:

* Age > 18 years
* Patients with postdural puncture headache defined as moderate to severe postural headache (VAS >= 30mm) after lumbar puncture or accidental dural puncture during epidural insertion with an onset within 3 days following the puncture.
* Lack of headache remission within 1 day after dural puncture and after treatment with fluids, caffeine and paracetamol
* Patients who have given their written informed consent for participation in the study after fully understanding the protocol content and limitations.

Exclusion Criteria:

* Patients who cannot cooperate to the study
* Patients who does not understand or speak Danish
* Allergy to the drugs used in the study
* Has taken opioids within 12 hours prior to intervention

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients who were included in main study NCT03652714
Sampling Method: Non-Probability Sample
Enrollment: 38 (Actual)
Dates: Start 2021-11-26 (Actual); Primary Completion 2022-04-19 (Actual); Study Completion 2022-04-19 (Actual)

PRIMARY OUTCOMES:
Migraine Disability Assessment Test score | 3 months following initial block
  Disability due to headache defined as moderate to severe disability measured with Migraine Disability Assessment Test Score (MIDAS) ranging from no disability at a score of 0 to severe disability at a score of 21+
Average pain score | 3 months following initial block
  Average pain score measured on a 0-10 pain rating scale (VAS) with 0 meaning no pain and 10 being the worst pain imaginable.

SECONDARY OUTCOMES:
Migraine Disability Assessment Test score | 3 previous months
  Disability due to headache is defined as moderate to severe disability measured with Migraine Disability Assessment Test Score (MIDAS) ranging from no disability at a score of 0 to severe disability at a score of 21+
Average pain score | 3 previous months
  Average pain score measured on a 0-10 pain rating scale (VAS) with 0 meaning no pain and 10 being the worst pain imaginable.
Days with headache | 3 months following initial block as well as the last 3 months
  Number of days with headache
Short term side effects | From date of initial block application until time of questionaire and inclusion in follow up study, assessed up to 60 months.
  Side effects following the block are defined as side effects with a duration of less than 3 months
Long term side effects | From date of initial block application until time of questionaire and inclusion in follow up study, assessed up to 60 months.
  Side effects following the block defined as side effects with a duration of more than 3 months

CONTACTS AND LOCATIONS:
Locations (1):
- Bispebjerg and Frederiksberg Hospital, University of Copenhagen, Copenhagen, Denmark